CLINICAL TRIAL: NCT01664598
Title: A Multicenter, Open-label, Single Arm, Long Term Extension Study of WA19926 to Describe Safety During Treatment With Tocilizumab in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: An Extension Study of WA19926 of the Long-Term Safety of Tocilizumab (RoActemra/Actemra) in Patients With Early Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28124
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental)
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 8 mg/kg administered intravenously (IV) every 4 weeks for 104 weeks
  Other Names: RoActemra; Actemra

SUMMARY:
This open-label, single arm, multicenter long-term extension study of WA19926 evaluated the safety and efficacy of tocilizumab (RoActemra/Actemra) in participants with moderate to severe rheumatoid arthritis who completed the 104-week WA19926 core study. Eligible patients received tocilizumab 8 mg/kg intravenously every 4 weeks for up to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants who complete their last WA19926 core study visit (Week 104) and who may benefit from study drug treatment according to the Investigator's assessment
* No current or recent adverse event or laboratory finding preventing the use of the study drug dose of RoActemra/Actemra 8 mg/kg at baseline visit
* Women of childbearing potential must agree to use adequate contraception as defined by protocol during the treatment period

Exclusion Criteria:

* Pregnant females
* Participants who have withdrawn prematurely from the WA19926 core study for any reason
* Treatment with any investigational agent or cell-depleting therapies since the last administration of study drug in WA19926
* Treatment with an anti-tumor necrosis factor (TNF) or anti-interleukin (IL) 1 agent, or a T-cell costimulation modulator since the last administration of study drug in WA19926
* Immunization with a live/attenuated vaccine since the last administration of study drug in WA19926
* Diagnosis since last WA19926 visit (Week 104) of rheumatic autoimmune disease other than rheumatoid arthritis
* Diagnosis since last WA19926 visit (Week 104) of inflammatory joint disease other than rheumatoid arthritis
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, including tocilizumab and its excipients
* Evidence of severe uncontrolled concomitant disease or disorder
* Known active or history of recurrent infections
* Active tuberculosis requiring treatment in the previous 3 years
* History of alcohol, drug or chemical abuse since inclusion in the WA19926 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Russia (8):
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Tula
  - Voronezh
  - Yaroslavl
  - Yekaterinburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the 104-week core study WA19926 and could benefit from tocilizumab treatment based on the Investigator's judgment were enrolled in this study.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 49
Completed | 43
Not Completed | 6
Not completed — Sponsor Decision | 1
Not completed — Withdrawal of Informed Consent | 4
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS), includes all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a study participant given administered a pharmaceutical product, regardless of the cause of the AE. A SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant. AESIs included serious infections (including opportunistic infections) and abnormal liver function tests.
Time Frame: Up to 112 weeks
Population: Full Analysis Set (FAS) included all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants
  Adverse Events | 69.4
  SAEs | 10.2
  AESIs | 17.2

2. Primary Outcome: Percentage of Adverse Events (AEs) Leading to Dose Modification and AEs Leading to Study Withdrawal
Description: An AE is any untoward medical occurrence in a study participant given administered a pharmaceutical product, regardless of the cause of the AE.
Time Frame: Up to 112 weeks
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Measure: Number; unit: percentage of adverse events
Units Other Than Participants: adverse events
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
Number analyzed (adverse events) | 87
percentage of adverse events
  AEs Leading to Dose Modification | 34.5
  AEs Leading to Study Withdrawal | 1.1

3. Primary Outcome: Percentage of Adverse Events With Severity as Mild, Moderate, and Severe
Time Frame: Up to 112 weeks
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Measure: Number; unit: percentage of adverse events
Units Other Than Participants: adverse events
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
Number analyzed (adverse events) | 87
percentage of adverse events
  Mild | 62.1
  Moderate | 36.8
  Severe | 1.1

4. Secondary Outcome: Percent Change From Baseline in the Disease Activity Index 28 Erythrocyte Sedimentation Rate (DAS28-ESR) Over Time
Description: The DAS28-ESR Scale is a measure of a participant's disease activity. It is based on tender joint count (28 joints), swollen joint count (28 joints), a participant's assessment of disease activity, and erythrocyte sedimentation rate. DAS28-ESR is expressed as a score on a scale with a minimum score of 0 (low disease activity ) to a maximum score of 10 (high disease activity). A negative mean percent change from baseline indicates a decrease in disease activity, and a positive mean percent change from baseline indicates an increase in disease activity.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab. Here, number of participants analyzed is the total participants who were evaluable for this outcome measure, and 'n' is the total number of participants who were evaluated at a specific time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 42
percent change
  Change at Week 12 (n=42) | -35.4 (30.4)
  Change at Week 24 (n=40): number analyzed (Participants) | 40
  Change at Week 24 (n=40) | -27.2 (35.4)
  Change at Week 36 (n=39): number analyzed (Participants) | 39
  Change at Week 36 (n=39) | -29.3 (48.4)
  Change at Week 48 (n=33): number analyzed (Participants) | 33
  Change at Week 48 (n=33) | -24.6 (41.0)
  Change at Week 56 (n=34): number analyzed (Participants) | 34
  Change at Week 56 (n=34) | -32.5 (31.9)
  Change at Week 68 (n=32): number analyzed (Participants) | 32
  Change at Week 68 (n=32) | -38.3 (25.6)
  Change at Week 80 (n=28): number analyzed (Participants) | 28
  Change at Week 80 (n=28) | -29.4 (33.5)
  Change at Week 92 (n=22): number analyzed (Participants) | 22
  Change at Week 92 (n=22) | -26.9 (30.9)
  Change at Week 104 (n=26): number analyzed (Participants) | 26
  Change at Week 104 (n=26) | -38.1 (25.9)

5. Secondary Outcome: Percent Change From Baseline in the Simplified Disease Activity Index (SDAI) Over Time
Description: The Simplified Disease Activity Index (SDAI) is the numerical sum of five outcome parameters: tender joint count (TJC) and swollen joint count (SJC), based on a 28-joint assessment, patient and physician global assessment assessed on 0-10 centimeter (cm) visual analogue scale (VAS), where 0 = no disease activity and 10 = worst disease activity, and level of C-reactive protein (CRP, mg/dL). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high (or severe) disease activity. A negative mean percent change from baseline indicates a decrease in disease activity, and a positive mean percent change from baseline indicates an increase in disease activity.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 38
percent change
  Change at Week 12 (n=37): number analyzed (Participants) | 37
  Change at Week 12 (n=37) | -45.5 (33.9)
  Change at Week 24 (n=36): number analyzed (Participants) | 36
  Change at Week 24 (n=36) | -34.7 (45.6)
  Change at Week 36 (n=38) | -6.3 (221.1)
  Change at Week 48 (n=36): number analyzed (Participants) | 36
  Change at Week 48 (n=36) | -12.4 (84.3)
  Change at Week 56 (n=34): number analyzed (Participants) | 34
  Change at Week 56 (n=34) | -39.3 (66.4)
  Change at Week 68 (n=35): number analyzed (Participants) | 35
  Change at Week 68 (n=35) | -47.3 (39.6)
  Change at Week 80 (n=36): number analyzed (Participants) | 36
  Change at Week 80 (n=36) | -30.3 (66.9)
  Change at Week 92 (n=36): number analyzed (Participants) | 36
  Change at Week 92 (n=36) | -12.5 (140.1)
  Change at Week 104 (n=35): number analyzed (Participants) | 35
  Change at Week 104 (n=35) | -28.8 (115.7)

6. Secondary Outcome: Change From Baseline in Tender Joint Count 66 (TJC 66) Over Time
Description: Number of tender joints was determined by examination of 66 joints, as assessed through pressure and passive joint motion during physical examination.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab. Here, 'n' is the total number of participants who were evaluated at a specific time point.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
tender joints
  Change at Week 12 (n=49) | -5.0 (6.7)
  Change at Week 24 (n=47): number analyzed (Participants) | 47
  Change at Week 24 (n=47) | -5.7 (9.5)
  Change at Week 36 (n=47): number analyzed (Participants) | 47
  Change at Week 36 (n=47) | -6.6 (10.4)
  Change at Week 48 (n=46): number analyzed (Participants) | 46
  Change at Week 48 (n=46) | -6.2 (11.8)
  Change at Week 56 (n=44): number analyzed (Participants) | 44
  Change at Week 56 (n=44) | -6.7 (10.6)
  Change at Week 68 (n=45): number analyzed (Participants) | 45
  Change at Week 68 (n=45) | -6.6 (10.6)
  Change at Week 80 (n=45): number analyzed (Participants) | 45
  Change at Week 80 (n=45) | -6.2 (10.8)
  Change at Week 92 (n=43): number analyzed (Participants) | 43
  Change at Week 92 (n=43) | -6.3 (11.9)
  Change at Week 104 (n=43): number analyzed (Participants) | 43
  Change at Week 104 (n=43) | -7.4 (10.9)

7. Secondary Outcome: Change From Baseline in Swollen Joint Count 66 (SJC 66) Over Time
Description: Number of swollen joints was determined by examination of 66 joints, as assessed through pressure and passive joint motion during physical examination.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
swollen joints
  Change at Week 12 (n=49) | -3.5 (7.9)
  Change at Week 24 (n=47): number analyzed (Participants) | 47
  Change at Week 24 (n=47) | -3.7 (8.2)
  Change at Week 36 (n=47): number analyzed (Participants) | 47
  Change at Week 36 (n=47) | -4.5 (9.9)
  Change at Week 48 (n=46): number analyzed (Participants) | 46
  Change at Week 48 (n=46) | -4.6 (9.9)
  Change at Week 56 (n=44): number analyzed (Participants) | 44
  Change at Week 56 (n=44) | -4.7 (9.7)
  Change at Week 68 (n=45): number analyzed (Participants) | 45
  Change at Week 68 (n=45) | -4.9 (9.7)
  Change at Week 80 (n=45): number analyzed (Participants) | 45
  Change at Week 80 (n=45) | -4.6 (9.7)
  Change at Week 92 (n=43): number analyzed (Participants) | 43
  Change at Week 92 (n=43) | -4.3 (10.2)
  Change at Week 104 (n=43): number analyzed (Participants) | 43
  Change at Week 104 (n=43) | -5.0 (10.0)

8. Secondary Outcome: Percentage of Participants With Treatment-Free Remission According to DAS28-ESR/SDAI Remission Criteria
Description: Treatment-free remission is remission at two consecutive assessment visits (every 12 weeks) after discontinuing study drug on the second assessment visit. Clinical remission is DAS28-ESR score <2.6 and/or SDAI score ≤3.3. The DAS28-ESR scale is a measure of a participant's disease activity based on tender joint count (28 joints), swollen joint count (28 joints), a participant's assessment of disease activity, and ESR. DAS28-ESR scored on a scale with a minimum score of 0 (low disease activity) to a maximum score of 10 (high disease activity). The SDAI is sum of TJC and SJC, based on a 28-joint assessment, patient and physician global assessment assessed on 0-10 centimeter visual analogue scale (VAS), where 0 = no disease activity and 10 = worst disease activity, and level of C-reactive protein (CRP, mg/dL). SDAI total score = 0-86. SDAI <=3.3 indicates clinical remission, >3.4 to 11=low disease activity, >11 to 26=moderate disease activity, and >26=high (or severe) disease activity.
Time Frame: Up to 104 weeks
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percentage of participants | 71.4

9. Secondary Outcome: Time to Rheumatoid Arthritis Recurrence in Participants Who Achieved Treatment-Free Remission
Description: Time to rheumatoid arthritis (RA) recurrence = period from treatment-free remission to RA recurrence. RA recurrence was worsening of disease activity with treatment beyond supportive therapy.
Time Frame: Up to 104 weeks
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab. Analysis was performed on those participants who achieved treatment-free remission.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Tocilizumab
Number analyzed (Participants) | 35
weeks | 23 [17.6 to 28.4]

10. Secondary Outcome: Percent Change in Participant's General Assessment of Disease Activity (Severity of Disease) VAS Over Time
Description: The participant's overall assessment of their current disease activity was displayed on a 100-millimeter (mm) horizontal VAS. The left-hand extreme (0 mm) of the line was described as "no disease activity" (symptom free and no arthritis symptoms) and the right-hand extreme (100 mm) was described as "maximum disease activity" (maximum arthritis disease activity). The change in Patient Global Assessment of Disease Activity was determined as the difference in values from baseline at each visit.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: FAS included all randomized participants enrolled in the study who received at least one dose of tocilizumab. Here, number of participants analyzed is the total participants who were evaluable for this outcome measure and 'n' is the total number of participants who were evaluated at specific time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percent change
  Change at Week 12 (n=48): number analyzed (Participants) | 48
  Change at Week 12 (n=48) | -19.6 (45.7)
  Change at Week 24 (n=46): number analyzed (Participants) | 46
  Change at Week 24 (n=46) | -20.3 (49.8)
  Change at Week 36 (n=46): number analyzed (Participants) | 46
  Change at Week 36 (n=46) | -17.5 (60.6)
  Change at Week 48 (n=45): number analyzed (Participants) | 45
  Change at Week 48 (n=45) | 6.1 (92.8)
  Change at Week 56 (n=43): number analyzed (Participants) | 43
  Change at Week 56 (n=43) | -14.2 (63.8)
  Change at Week 68 (n=44): number analyzed (Participants) | 44
  Change at Week 68 (n=44) | -19.3 (48.6)
  Change at Week 80 (n=44): number analyzed (Participants) | 44
  Change at Week 80 (n=44) | -9.2 (58.1)
  Change at Week 92 (n=43): number analyzed (Participants) | 43
  Change at Week 92 (n=43) | -4.7 (67.2)
  Change at Week 104 (n=42): number analyzed (Participants) | 42
  Change at Week 104 (n=42) | -14.2 (75.7)

11. Secondary Outcome: Percent Change in Participant's Assessment of Pain (VAS) Over Time
Description: Participants' pain was assessed using a 10-mm horizontal VAS (0 to 10 mm) where 0=pain absent and 10=intolerable pain. Participants responded by placing a mark on the line to indicate their current level of pain; the distance from the left edge to the mark was recorded.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
percent change
  Change at Week 12 (n=48): number analyzed (Participants) | 48
  Change at Week 12 (n=48) | -21.8 (43.2)
  Change at Week 24 (n=46): number analyzed (Participants) | 46
  Change at Week 24 (n=46) | -20.3 (44.9)
  Change at Week 36 (n=46): number analyzed (Participants) | 46
  Change at Week 36 (n=46) | -25.4 (50.0)
  Change at Week 48 (n=45): number analyzed (Participants) | 45
  Change at Week 48 (n=45) | 4 (131.4)
  Change at Week 56 (n=43): number analyzed (Participants) | 43
  Change at Week 56 (n=43) | -19.8 (66.3)
  Change at Week 68 (n=44): number analyzed (Participants) | 44
  Change at Week 68 (n=44) | -19.9 (57.6)
  Change at Week 80 (n=44): number analyzed (Participants) | 44
  Change at Week 80 (n=44) | -17.1 (54.2)
  Change at Week 92 (n=43): number analyzed (Participants) | 43
  Change at Week 92 (n=43) | -10.9 (59.2)
  Change at Week 104 (n=42): number analyzed (Participants) | 42
  Change at Week 104 (n=42) | -20.5 (61.3)

12. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire (HAQ-DI) Score Over Time
Description: The HAQ-DI was used to assess the physical ability and functional status of participants as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from 4 response categories, ranging from 'without any difficulty' (Score=0) to 'unable to do' (Score=3). The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 56, 68, 80, 92 and 104
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 49
score on a scale
  Change at Week 12 (n=49) | -0.2 (0.4)
  Change at Week 24 (n=46): number analyzed (Participants) | 46
  Change at Week 24 (n=46) | -0.2 (0.4)
  Change at Week 36 (n=46): number analyzed (Participants) | 46
  Change at Week 36 (n=46) | -0.1 (0.4)
  Change at Week 48 (n=45): number analyzed (Participants) | 45
  Change at Week 48 (n=45) | 0.0 (0.5)
  Change at Week 56 (n=44): number analyzed (Participants) | 44
  Change at Week 56 (n=44) | -0.1 (0.6)
  Change at Week 68 (n=45): number analyzed (Participants) | 45
  Change at Week 68 (n=45) | -0.2 (0.5)
  Change at Week 80 (n=45): number analyzed (Participants) | 45
  Change at Week 80 (n=45) | -0.2 (0.5)
  Change at Week 92 (n=43): number analyzed (Participants) | 43
  Change at Week 92 (n=43) | 0.0 (0.6)
  Change at Week 104 (n=43): number analyzed (Participants) | 43
  Change at Week 104 (n=43) | -0.1 (0.5)

ADVERSE EVENTS:
Time Frame: Up to 112 Weeks
Description: FAS includes all randomized participants enrolled in the study who received at least one dose of tocilizumab.
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 5/49
Other Adverse Events (participants affected / at risk) | 22/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=49)
Arrhythmia (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Jaw abscess (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=49)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 9
Bronchitis (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Dyslipidaemia (Metabolism and nutrition disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.